CLINICAL TRIAL: NCT00948870
Title: Trial of Chinese Prescription Shugan Decoction on Irritable Bowel Syndrome（Diarrhea Type）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHTCM-002
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2009-08

CONDITIONS: Irritable Bowel Syndrome; Traditional Chinese Medicine
Keywords: alternative medicine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — shugan liangxue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shugan Decoction (Experimental)
  Interventions: Drug: Shugan decoction
- low does of Shugan decoction (Placebo Comparator)
  Interventions: Drug: Shugan decoction

INTERVENTIONS:
Drug: Shugan decoction — Decoction ,two times a day,one bag of decoction one time

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the Chinese prescription Shugan decoction on irritable bowel syndrome（diarrhea type）.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of irritable bowel syndrome（diarrhea type）
* Male of female patients between 18-65 years old
* Written informed consent

Exclusion Criteria:

* Discrepancy of irritable bowel syndrome
* Diarrhea-type of irritable bowel syndrome combine with intestinal disease
* Combined with severe heart, gallbladder, kidney, endocrine system, hemopoietic system or nervous system disease.
* Pregnancy or breast feeding women, or unwilling to have contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Symptoms and conditions of tongue and pulse | 4 weeks

SECONDARY OUTCOMES:
Indicates of liver and renal function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xie Jianqun, Phd, Study Director — Shanghai University of Chinese Medicine
Locations (1):
- Longhua hospital, Shanghai, Shanghai Municipality, China